CLINICAL TRIAL: NCT01781247
Title: MI-SPRINT (Myocardial Infarction - Stress PRevention INTervention): A Randomized Controlled Minimal Early Behavioral Intervention Trial to Reduce the Development of Posttraumatic Stress Caused by Acute Myocardial Infarction
Brief Title: Myocardial Infarction - Stress Prevention Intervention
Acronym: MI-SPRINT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Population of eligible patients smaller than anticipated
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); University of Bern (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 170/12; 140960 (Other Grant/Funding Number: SNF); 2258 (Other: Bern University Hospital)
Record Dates: First submitted 2013-01-21; First posted 2013-01-31 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Stress Disorders, Post-Traumatic; Myocardial Infarction
Keywords: Stress Disorders, Post-Traumatic; Myocardial Infarction; Psychotherapy; Preventive Therapy; Randomized Controlled Trial; Cardiovascular Diseases; Psychological Stress; Biomarkers
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Myocardial Infarction; Cardiovascular Diseases; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will participate in one single counseling session of 45 minutes (the minimal behavioral intervention) that targets specific MI-triggered traumatic reactions.
  Interventions: Behavioral: Minimal behavioral intervention
- Control group (Active Comparator): Patients in the control group will participate in one single counseling session of 45 minutes (the control intervention) that targets more general information about the role of psychological stress in coronary heart disease.
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Behavioral: Minimal behavioral intervention — The minimal behavioral intervention consists of one single counseling session of 45 minutes that targets specific MI-triggered traumatic reactions. The focus of the intervention is an educational and resource-oriented approach targeting individual patient resources and cognitive (re)structuring.
  Arms: Intervention group
Behavioral: Control intervention — The control intervention consists of one single counseling session of 45 minutes that targets more general information about the role of psychological stress in coronary heart disease. Any terminology related to "trauma" will be completely avoided.
  Arms: Control group

SUMMARY:
Posttraumatic Stress Disorder (PTSD) is a mental disorder that may occur after someone experiences a traumatic event. Between 10-20% of patients may develop PTSD in response to the traumatic experience of myocardial infarction (MI). PTSD is associated with impaired quality of life, social functioning, and high economic burden to the society. Posttraumatic stress attributable to MI has also been shown to be predictive of poor cardiovascular prognosis, whereby this link might relate to several atherothrombotic processes. Therefore the prevention of PTSD after MI is of high relevance. Guidelines have been published for early interventions to prevent the development of posttraumatic stress after different types of trauma but not in terms of acute MI as a traumatic event.

The overarching aim of the planned trial is to test whether a minimal behavioral intervention performed shortly after acute MI in patients at a high risk to develop PTSD and in the setting of a coronary care unit reduces the development of posttraumatic stress.

The primary hypothesis is that posttraumatic stress levels at the 3-month follow-up will be at least 20% lower in the intervention group than in the control group, and that this effect will last up to 12 months after the intervention. The secondary hypothesis is that the intervention group will show better psychosocial functioning, and a more favourable cardiometabolic biomarker profile than the control group 3 and 12 month after the intervention.

DETAILED DESCRIPTION:
Background

Posttraumatic Stress Disorder (PTSD) is a mental disorder that may occur after someone experiences a traumatic event. Between 10-20% of patients may develop PTSD in response to the traumatic experience of myocardial infarction (MI). Sociodemographic and psychosocial variables, including perceived distress during MI, have been identified as "risk factors" for the development of posttraumatic stress in the aftermath of MI. PTSD is associated with impaired quality of life, social functioning, and high economic burden to the society. Posttraumatic stress attributable to MI has also been shown to be predictive of poor cardiovascular prognosis, whereby this link might relate to atherothrombotic processes like endothelial dysfunction, dyslipidemia, inflammation, and coagulation. Therefore the prevention of PTSD after MI is of high relevance. Guidelines have been published for early interventions to prevent the development of posttraumatic stress after different types of trauma. A recent systematic review and meta-analysis on randomized controlled trials of early psychological interventions designed to prevent symptoms of PTSD found a benefit, but only if treatment was provided to symptomatic individuals and trauma-focused. The impact of such an intervention on posttraumatic stress in response to a myocardial infarction has not been assessed so far. The planned project is the first to test, if the development of posttraumatic stress can successfully be prevented in MI patients at high risk to develop PTSD through a minimal behavioral intervention that is feasible.

Objective

Primary aim: The overarching aim of the planned project is to investigate in a randomized-controlled trial whether a minimal (single counseling session of 45 minutes plus an information booklet) and early-on (within 48 hours after myocardial infarction) administered behavioral intervention reduces the development of clinician-rated posttraumatic stress levels attributable to MI in patients at a high risk to develop clinically relevant levels of posttraumatic stress.

Secondary aim: A further aim is to investigate whether the behavioral intervention improves psychosocial functioning and favorably affects cardiometabolic risk markers.

Methods

Patients considered to be at "high risk" to develop posttraumatic stress will be randomized to one single counseling session of 45 minutes (either targeting specific MI-triggered traumatic reactions or more general information about the role of psychological stress in coronary heart disease). The session will be performed by the study therapist in the coronary care unit within 48 hours after the patient has reached stable circulatory condition. Each patient will additionally receive written study material in the form of an information booklet. Medical variables, sociodemographic factors and cardiometabolic biomarkers will also be determined.

At 3-month and 12-month follow-up each patient will be assessed for interviewer-rated posttraumatic stress levels, psychosocial functioning, and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* STEMI (ST-elevated myocardial infarction) or non-STEMI
* Stable circulatory condition
* Numeric Rating Scale (NRS) (0-10): a score of at least 5 for "pain (during MI)" plus a score of at least 5 for "fear of dying (until admission to the CCU)" and/or "making sorrows and feeling helpless (when being told about having MI)"
* Written informed consent

Exclusion Criteria

* Participating in any other randomized-controlled trial run by the Cardiology Department of the University Hospital of Bern
* Emergency coronary artery bypass graft surgery
* Comorbid serious disease likely to cause death within 1 year
* Current clinically severe depression
* Not fully oriented to the situation, person, and place
* Cognitive impairment according to an adapted short version of the Mini-Mental State Examination
* Insufficient knowledge of German language in reading and understanding
* Affirmation of suicidal ideation in the last two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinician-rated posttraumatic stress level | 3 months
  Measured by Clinician-Administered PTSD Scale (CAPS) (German version)

SECONDARY OUTCOMES:
Clinician-rated posttraumatic stress level | 12 months
  Measured by Clinician-Administered PTSD Scale (CAPS) (German version)
Self-rated Posttraumatic Stress | 3 and 12 months
  Measured by Posttraumatic Diagnostic Scale (PDS) (German version); The term "event" will be replaced with the term "heart attack" to assess MI-specific posttraumatic stress.
Quality of Life | 3 and 12 months
  Measured by EuroQol group 5 dimension questionnaire (EQ-5D) (German version)
Depressive Symptoms | 3 and 12 months
  Measured by Beck Depression Inventory (BDI) (German version)
Overall psychological distress | 3 and 12 months
  Measured by self-rated symptom checklist-9 (SCL-9-K) (German version)
Positive and Negative Affect | 3 and 12 months
  Measured by 20-item Global Mood Scale (GMS) (German version)
Time duration to recurrence at previous job (incl. part-time) | 3 and 12 months
Time duration to recurrence at household to extent at least 50% | 3 and 12 months
Vitality status | 3 and 12 months
  Measured if alive or deceased (with cause of death)
Recurrent Hospitalisations | 3 and 12 months
  Measured: number and cause
Recurrent Doctor Visits - general practitioner as well as specialist | 3 and 12 months
  Measured: number and cause
Inflammation Markers | 3 and 12 months
  Measured by high sensitive C-reactive protein, Interleukin-6, Tumor necrosis factor alpha, Interleukin-4
Hemostasis Markers | 3 and 12 months
  Measured by Fibrinogen, D-dimer, von Willebrand factor (antigen)
Metabolic Factors | 3 and 12 months
  Measured by total cholesterol, Low-density lipoprotein-Cholesterol, High-density lipoprotein-Cholesterol, triglycerides, glucose, HbA1c
Anthropometric measurements | 3 and 12 months
  Measured by weight, height, body mass index (kg/m2), waist circumference, hip circumference, waist-to-hip ratio
Resting hemodynamics | 3 and 12 months
  Measured by heart rate, systolic blood pressure, diastolic blood pressure
Heart rate variability | 3 and 12 months
  Measured by total power, high frequency power, low frequency power, low-to-high frequency power ratio
Stress Hormones | 3 and 12 months
  Measured by plasma cortisol, norepinephrine, epinephrine

CONTACTS AND LOCATIONS:
Overall Officials: Roland von Känel, Prof. Dr. med., Principal Investigator; Jean-Paul Schmid, PD Dr. med., Study Chair; Ulrich Schnyder, Prof. Dr. med., Study Chair; Hansjörg Znoj, Prof. Dr. phil., Study Chair; Jürgen Barth, PD Dr. phil., Study Chair
Locations (1):
- Dep. of General Internal Medicine, Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Gander ML, von Kanel R. Myocardial infarction and post-traumatic stress disorder: frequency, outcome, and atherosclerotic mechanisms. Eur J Cardiovasc Prev Rehabil. 2006 Apr;13(2):165-72. doi: 10.1097/01.hjr.0000214606.60995.46. PMID 16575268
- [Background] Edmondson D, Richardson S, Falzon L, Davidson KW, Mills MA, Neria Y. Posttraumatic stress disorder prevalence and risk of recurrence in acute coronary syndrome patients: a meta-analytic review. PLoS One. 2012;7(6):e38915. doi: 10.1371/journal.pone.0038915. Epub 2012 Jun 20. PMID 22745687
- [Background] von Kanel R, Hari R, Schmid JP, Wiedemar L, Guler E, Barth J, Saner H, Schnyder U, Begre S. Non-fatal cardiovascular outcome in patients with posttraumatic stress symptoms caused by myocardial infarction. J Cardiol. 2011 Jul;58(1):61-8. doi: 10.1016/j.jjcc.2011.02.007. Epub 2011 Apr 13. PMID 21493042
- [Background] Roberts NP, Kitchiner NJ, Kenardy J, Bisson JI. Systematic review and meta-analysis of multiple-session early interventions following traumatic events. Am J Psychiatry. 2009 Mar;166(3):293-301. doi: 10.1176/appi.ajp.2008.08040590. Epub 2009 Feb 2. PMID 19188285
- [Background] Ehlers A, Clark DM, Hackmann A, McManus F, Fennell M, Herbert C, Mayou R. A randomized controlled trial of cognitive therapy, a self-help booklet, and repeated assessments as early interventions for posttraumatic stress disorder. Arch Gen Psychiatry. 2003 Oct;60(10):1024-32. doi: 10.1001/archpsyc.60.10.1024. PMID 14557148
- [Derived] von Kanel R, Meister-Langraf RE, Zuccarella-Hackl C, Znoj H, Pazhenkottil AP, Schmid JP, Barth J, Schnyder U, Princip M. Association Between Changes in Post-hospital Cardiac Symptoms and Changes in Acute Coronary Syndrome-Induced Symptoms of Post-traumatic Stress. Front Cardiovasc Med. 2022 Apr 14;9:852710. doi: 10.3389/fcvm.2022.852710. eCollection 2022. PMID 35498017
- [Derived] von Kanel R, Meister-Langraf RE, Pazhenkottil AP, Barth J, Schnyder U, Schmid JP, Znoj H, Princip M. Insomnia Symptoms and Acute Coronary Syndrome-Induced Posttraumatic Stress Symptoms: A Comprehensive Analysis of Cross-sectional and Prospective Associations. Ann Behav Med. 2021 Oct 4;55(10):1019-1030. doi: 10.1093/abm/kaaa128. PMID 33580657
- [Derived] von Kanel R, Schmid JP, Meister-Langraf RE, Barth J, Znoj H, Schnyder U, Princip M, Pazhenkottil AP. Pharmacotherapy in the Management of Anxiety and Pain During Acute Coronary Syndromes and the Risk of Developing Symptoms of Posttraumatic Stress Disorder. J Am Heart Assoc. 2021 Jan 19;10(2):e018762. doi: 10.1161/JAHA.120.018762. Epub 2021 Jan 12. PMID 33432839
- [Derived] von Kanel R, Princip M, Schmid JP, Barth J, Znoj H, Schnyder U, Meister-Langraf RE. Association of sleep problems with neuroendocrine hormones and coagulation factors in patients with acute myocardial infarction. BMC Cardiovasc Disord. 2018 Nov 21;18(1):213. doi: 10.1186/s12872-018-0947-5. PMID 30463526
- [Derived] Meister R, Princip M, Schmid JP, Schnyder U, Barth J, Znoj H, Herbert C, von Kanel R. Myocardial Infarction - Stress PRevention INTervention (MI-SPRINT) to reduce the incidence of posttraumatic stress after acute myocardial infarction through trauma-focused psychological counseling: study protocol for a randomized controlled trial. Trials. 2013 Oct 11;14:329. doi: 10.1186/1745-6215-14-329. PMID 24119487